CLINICAL TRIAL: NCT00167882
Title: The Influence of 5-Aminosalicylates on Thiopurine Metabolite Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2005/28
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-08

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Crohn's disease; Ulcerative colitis; Inflammatory bowel disease; azathioprine; 6-mercaptopurine; 5-aminosalicylate; metabolism
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Mesalamine

INTERVENTIONS:
Drug: 5-aminosalicylate (Pentasa, Ferring)

SUMMARY:
The purpose of this study is to determine the influence of different 5-aminosalicylate concentrations on the metabolism of azathioprine or 6-mercaptopurine in patients with inflammatory bowel disease.

DETAILED DESCRIPTION:
Background:

The concomitant use of 5-aminosalicylates (5ASA) next to azathioprine (AZA) or 6-mercaptopurine (6MP) in the treatment of inflammatory bowel disease (IBD) may lead to an increased effectiveness of therapy as higher levels of the active metabolite of AZA/6MP (6-thioguaninenucleotides (6TGNs) are measured.

Objectives:

To determine the influence of 5-ASA compounds and its metabolites on the metabolites of AZA/6MP (6TGNs + 6-methylmercaptopurine (6MMP).

Methods:

Patients with quiescent disease under AZA/6MP therapy are eligible. Patients will receive three succeeding regimes (5ASA 2 gram/5ASA 4 gram/ no 5ASA) of 4 weeks next to the standard AZA/6MP therapy. At the start and at the end of every regime 5ASA and its major metabolite (N-acetyl-5ASA) will be determined in serum next to the measurement of 6TGNs and 6MMP in erythrocytes. The safety will monitored by standard laboratory parameters every four weeks.

Population:

Patients with IBD in remission and unchanged AZA/6MP dosages for at least 4 weeks.

Medication:

5ASA (Pentasa ® granules; Ferring) will be administered orally in dosages of 2 or 4 grams daily for a period of 4 weeks.

Endpoints:

The rise or decrease in 6TGNs and 6MMP during the different 5ASA regimes. The evaluation of the safety of co-administrating 5ASA next to AZA/6MP.

Risks:

Side effects of 5ASA use are limited and well known. Some case reports have described the potential risk of developing a myelodepression when AZA/6MP and 5ASA are given together due to the rise in 6TGNs. However, in daily practice both drugs are administered together frequently. The risks of the frequent blood draws are minimal and usually self-limiting (haematoma).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged between 18 - 70 years
* Informed consent
* Diagnosis of CD or UC for at least 6 months (histological and endoscopically confirmed)
* Steady state AZA of 6-MP use (an unchanged thiopurine regime for at least 4 weeks)
* Normal liver and kidney function (ALAT / AP / creatinin < 2 x upper normal limit)
* Quiescent disease (HBI score ≤ 4 for CD or modified TLWI score ≤ 4 for UC)

Exclusion Criteria:

* Bone marrow suppression (platelets / leucocytes < 1 x lower normal level)
* Presence of active infection (fever and CRP > 1 x upper normal limit)
* Anemia (hemoglobin < 6 mmol)
* Known duodenal Crohn's disease interfering significantly with resorptive area
* Small bowel surgery interfering significantly with resorptive area
* Known intolerance to 5-ASA compounds
* Current use of 5-ASA compounds
* Use of 5-ASA compounds within the last 30 days
* Concomitant use of allopurinol, ACE-inhibitors or furosemide
* Pregnancy, expected pregnancy or lactation within 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-07; Study Completion 2006-08

PRIMARY OUTCOMES:
To determine the influence of 5-ASA compounds and its metabolites on the 6-TGN level during steady state AZA or 6-MP dosages

SECONDARY OUTCOMES:
To determine the influence of 5-ASA compounds and its metabolites on the 6-MMP level during steady state AZA or 6-MP dose
To determine the influence of 5-ASA compounds and its metabolites on the 6-TGMP, 6-TGDP and 6-TGTP levels during steady state AZA or 6-MP dosages
To evaluate the safety of co-administrating 5-ASA and AZA or 6-MP in IBD patients

CONTACTS AND LOCATIONS:
Overall Officials: K.H.N. de Boer, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Maasland Hospital, Sittard, Netherlands

REFERENCES:
- [Background] Derijks LJ, Gilissen LP, Engels LG, Bos LP, Bus PJ, Lohman JJ, Curvers WL, Van Deventer SJ, Hommes DW, Hooymans PM. Pharmacokinetics of 6-mercaptopurine in patients with inflammatory bowel disease: implications for therapy. Ther Drug Monit. 2004 Jun;26(3):311-8. doi: 10.1097/00007691-200406000-00016. PMID 15167634
- [Background] de Boer NK, de Graaf P, Wilhelm AJ, Mulder CJ, van Bodegraven AA. On the limitation of 6-tioguaninenucleotide monitoring during tioguanine treatment. Aliment Pharmacol Ther. 2005 Sep 1;22(5):447-51. doi: 10.1111/j.1365-2036.2005.02581.x. PMID 16128683
- [Background] Al Hadithy AF, de Boer NK, Derijks LJ, Escher JC, Mulder CJ, Brouwers JR. Thiopurines in inflammatory bowel disease: pharmacogenetics, therapeutic drug monitoring and clinical recommendations. Dig Liver Dis. 2005 Apr;37(4):282-97. doi: 10.1016/j.dld.2004.09.029. PMID 15788214